CLINICAL TRIAL: NCT01086228
Title: XIENCE V/PROMUS Everolimus-Eluting Stent System Japan Post-marketing Surveillance Protocol
Brief Title: XIENCE V/PROMUS Everolimus-Eluting Stent System Post-marketing Surveillance Protocol for Japan
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-384
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2017-08

CONDITIONS: Angina; Chronic Coronary Occlusion; Stent Thrombosis; Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: Drug eluting stents; Stents; Angioplasty
MeSH Terms: conditions — Angina Pectoris; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- XIENCE V / PROMUS stent: Only the patients treated with the XIENCE V / PROMUS stent during the index procedure will be analyzed.
  Interventions: Device: XIENCE V / PROMUS stent

INTERVENTIONS:
Device: XIENCE V / PROMUS stent — Patients receiving XIENCE V stent(s) or PROMUS stent(s) during their index procedure.

SUMMARY:
The objectives of this post-marketing surveillance, conducted in Japan, is to know the frequency, type and degree of device malfunction, to assure the safety of the medical device, and to collect information on evaluation of the efficacy and safety.

DETAILED DESCRIPTION:
The surveillance is to be conducted in accordance with the Japanese Ministerial Ordinance concerning the Standards for Postmarketing Surveillance and Tests of Medical Devices.

ELIGIBILITY:
Inclusion Criteria:

* Only XIENCE V stent(s)or PROMUS stent(s) is (are) implanted in the coronary vasculature during the index procedure.

Exclusion Criteria:

* Neither XIENCE V stent(s) nor PROMUS stent(s) is (are) implanted in the coronary vasculature during the index procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Only patients in Japan, who are eligible to receive treatment for coronary arteries using the XIENCE V / PROMUS Everolimus-Eluting Stent System are to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2010 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Thompson, Study Director — Abbott Medical Devices
Locations (47):
- Japan (47):
  - Site Reference ID/Investigator# 104727, Aichi
  - Site Reference ID/Investigator# 113428, Aichi
  - Site Reference ID/Investigator# 115745, Aichi
  - Site Reference ID/Investigator# 104424, Chiba
  - Site Reference ID/Investigator# 113645, Chiba
  - Site Reference ID/Investigator# 105015, Ehime
  - Site Reference ID/Investigator# 105148, Fukuoka
  - Site Reference ID/Investigator# 105177, Fukuoka
  - Site Reference ID/Investigator# 104677, Gifu
  - Site Reference ID/Investigator# 104365, Gunma
  - Site Reference ID/Investigator# 105038, Hiroshima
  - Site Reference ID/Investigator# 105043, Hiroshima
  - Site Reference ID/Investigator# 104236, Hokkaido
  - Site Reference ID/Investigator# 105963, Hyōgo
  - Site Reference ID/Investigator# 104326, Ibaraki
  - Site Reference ID/Investigator# 104606, Ishikawa
  - Site Reference ID/Investigator# 104607, Ishikawa
  - Site Reference ID/Investigator# 104528, Kanagawa
  - Site Reference ID/Investigator# 104536, Kanagawa
  - Site Reference ID/Investigator#104563, Kanagawa
  - Site Reference ID/Investigator# 104837, Kyoto
  - Site Reference ID/Investigator# 104838, Kyoto
  - Site Reference ID/Investigator# 104843, Kyoto
  - Site Reference ID/Investigator# 104844, Kyoto
  - Site Reference ID/Investigator# 104850, Kyoto
  - Site Reference ID/Investigator# 104658, Nagano
  - Site Reference ID/Investigator# 104990, Nara
  - Site Reference ID/Investigator# 105027, Okayama
  - Site Reference ID/Investigator# 105296, Okinawa
  - Site Reference ID/Investigator# 104864, Osaka
  - Site Reference ID/Investigator# 104898, Osaka
  - Site Reference ID/Investigator# 104906, Osaka
  - Site Reference ID/Investigator# 114863, Osaka
  - Site Reference ID/Investigator# 104407, Saitama
  - Site Reference ID/Investigator# 106044, Saitama
  - Site Reference ID/Investigator# 104697, Shizuoka
  - Site Reference ID/Investigator# 104356, Tochigi
  - Site Reference ID/Investigator# 105092, Tokushima
  - Site Reference ID/Investigator# 104448, Tokyo
  - Site Reference ID/Investigator# 104454, Tokyo
  - Site Reference ID/Investigator# 104473, Tokyo
  - Site Reference ID/Investigator# 104497, Tokyo
  - Site Reference ID/Investigator# 104510, Tokyo
  - Site Reference ID/Investigator# 104514, Tokyo
  - Site Reference ID/Investigator#104481, Tokyo
  - Site Reference ID/Investigator # 104285, Yamagata
  - Site Reference ID/Investigator# 104294, Yamagata

REFERENCES:
- [Derived] Aoki J, Kozuma K, Awata M, Nanasato M, Shiode N, Tanabe K, Yamaguchi J, Kusano H, Nie H, Kimura T; XIEVCE V/PROMUS PMS Investigators. Five-year clinical outcomes of everolimus-eluting stents from the post marketing study of CoCr-EES (XIENCE V/PROMUS) in Japan. Cardiovasc Interv Ther. 2019 Jan;34(1):40-46. doi: 10.1007/s12928-018-0515-z. Epub 2018 Feb 26. PMID 29484580
- [Derived] Shiode N, Kozuma K, Aoki J, Awata M, Nanasato M, Tanabe K, Yamaguchi J, Kusano H, Nie H, Kimura T; XIEVCE V/Promus PMS Investigators. The impact of coronary calcification on angiographic and 3-year clinical outcomes of everolimus-eluting stents: results of a XIENCE V/PROMUS post-marketing surveillance study. Cardiovasc Interv Ther. 2018 Oct;33(4):313-320. doi: 10.1007/s12928-017-0484-7. Epub 2017 Jul 19. PMID 28726115
- [Derived] Aoki J, Kozuma K, Awata M, Nanasato M, Shiode N, Tanabe K, Yamaguchi J, Kusano H, Nie H, Kimura T; XIEVCE V/PROMUS PMS Investigators. Three-Year Clinical Outcomes of Everolimus-Eluting Stents From the Post-Marketing Surveillance Study of Cobalt-Chromium Everolimus-Eluting Stent (XIENCE V/PROMUS) in Japan. Circ J. 2016;80(4):906-12. doi: 10.1253/circj.CJ-15-1181. Epub 2016 Jan 27. PMID 26821583

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2010 patients were registered. Of which 1 patient was excluded from this analysis. Therefore, 2009 patients (1,159 patients treated with XIENCE V; 850 patients treated with PROMUS) were included in the analysis.
Pre-assignment Details: Study has excluded those patients who were treated with stents other than CoCr-EES (XIENCE V or PROMUS), or underwent concomitant treatment of a graft vessel. Patients were invited to enroll in the study after apparently successful per-cutaneous coronary intervention (PCI).
Period: 8 Month Follow-up
Arm/Group | XIENCE V / PROMUS Stent
Started | 2009 (Analysis population)
Completed | 1938
Not Completed | 71
Period: 1-year Follow-up
Arm/Group | XIENCE V / PROMUS Stent
Started | 1938
Completed | 1894
Not Completed | 44
Period: 2-year Follow-up
Arm/Group | XIENCE V / PROMUS Stent
Started | 1894
Completed | 1834
Not Completed | 60
Period: 3-year Follow-up
Arm/Group | XIENCE V / PROMUS Stent
Started | 1834
Completed | 1767
Not Completed | 67
Period: 4-year Follow-up
Arm/Group | XIENCE V / PROMUS Stent
Started | 1767
Completed | 1664
Not Completed | 103
Period: 5-year Follow-up
Arm/Group | XIENCE V / PROMUS Stent
Started | 1664
Completed | 1012
Not Completed | 652

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analyzed for 2,009 patients (XIENCE V:1,159 ; PROMUS : 850).
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 2009
Age, Continuous [Median (Standard Deviation); unit: years] | 70.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 481
  Male | 1528
Region of Enrollment [Number; unit: participants]
  Japan | 2009

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stent Thrombosis (ST) as Per ARC Definition
Description: Definite ST occurred by either angiographic/pathologic confirmation of ST.
  Angiographic confirmation:The presence of a thrombus that originates in the stent/in the segment 5mm proximal/distal to the stent&presence of at least 1 of the following criteria within 48-hours:
  * Acute onset of ischemic symptoms at rest
  * New ischemic ECG changes
  * Typical rise&fall in cardiac biomarkers
  * Non-occlusive &occlusive thrombus
  Pathological confirmation:Evidence of recent thrombus within the stent determined at autopsy/via examination of tissue retrieved following thrombectomy.
  Probable ST may occur due to:
  * Unexplained death within first 30 days
  * Irrespective of the time after the index procedure,any MI that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of ST&in the absence of any other obvious cause.
  Possible ST occurred with any unexplained death from 30 days after intracoronary stenting until end of trial follow-up
Time Frame: Post Procedure to 1 Year
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 2009
participants
  Definite Stent Thrombosis | 6
  Probable Stent Thrombosis | 2
  Possible Stent Thrombosis | 6

2. Primary Outcome: Number of Participants With Stent Thrombosis (ST) as Per ARC Definition
Description: as for outcome 1
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1894
participants
  Definite Stent Thrombosis | 0
  Probable Stent Thrombosis | 0
  Possible Stent Thrombosis | 5

3. Primary Outcome: Number of Participants With Stent Thrombosis (ST) as Per ARC Definition
Description: as for outcome 1
Time Frame: From 2 years to 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1834
participants
  Definite Stent Thrombosis | 0
  Probable Stent Thrombosis | 0
  Possible Stent Thrombosis | 4

4. Secondary Outcome: Number of Participants With Adverse Events Related to Anti-platelet Medication
Time Frame: From post-procedure to 1 year
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 2009
participants
  Abnormal Non-Cardiac Lab Value/Test | 13
  Allergic Reaction | 10
  Bleeding | 32
  Cardiac | 3
  Cancer/Tumor | 0
  Gastro-intestinal | 4
  General/Musculoskeletal/Connective | 7
  Genito-urinary and renal disorder | 0
  Neurological/Psychiatric disorders | 3
  Vascular | 4

5. Secondary Outcome: Number of Participants With Adverse Events Related to Anti-platelet Medication
Time Frame: From 1 year to 2 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1894
participants
  Abnormal Non-Cardiac Lab Value/Test | 2
  Allergic Reaction | 0
  Bleeding | 5
  Cardiac | 0
  Cancer/Tumor | 1
  Gastro-intestinal | 0
  General/Musculoskeletal/Connective | 0
  Genito-urinary and renal disorder | 1
  Neurological/Psychiatric disorders | 0
  Vascular | 0

6. Secondary Outcome: Number of Participants With Adverse Events Related to Anti-platelet Medication
Time Frame: From 2 years to 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1834
participants
  Abnormal Non-Cardiac Lab Value/Test | 2
  Allergic Reaction | 0
  Bleeding | 3
  Cardiac | 1
  Cancer/Tumor | 0
  Gastro-intestinal | 0
  General/Musculoskeletal/Connective | 0
  Genito-urinary and renal disorder | 0
  Neurological/Psychiatric disorders | 1
  Vascular | 0

7. Secondary Outcome: Number of Participants With Adverse Events Related to Anti-platelet Medication
Time Frame: From 3 years to 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1767
participants
  Abnormal Non-Cardiac Lab Value/Test | 0
  Allergic Reaction | 0
  Bleeding | 9
  Cardiac | 0
  Cancer/Tumor | 0
  Gastro-intestinal | 0
  General/Musculoskeletal/Connective | 1
  Genito-urinary and renal disorder | 0
  Neurological/Psychiatric disorders | 1
  Vascular | 2

8. Secondary Outcome: Number of Participants With Adverse Events Related to Anti-platelet Medication
Time Frame: From 4 years to 5 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1664
participants
  Abnormal Non-Cardiac Lab Value/Test | 0
  Allergic Reaction | 0
  Bleeding | 3
  Cardiac | 0
  Cancer/Tumor | 0
  Gastro-intestinal | 2
  General/Musculoskeletal/Connective | 2
  Genito-urinary and renal disorder | 1
  Neurological/Psychiatric disorders | 1
  Vascular | 0

9. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: Percent Diameter Stenosis is defined as the value calculated as 100 * (1 - Minimum Luminal Diameter (MLD)/Reference vessel diameter (RVD)) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
Time Frame: Baseline
Population: Pre-procedure and immediate post-procedure angiograms were available from all of the analysis population of 2,009 patients (2,647 lesions), of which 1,850 lesions in 1548 patients were assessed by the core laboratory.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: lesions
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1548
Number analyzed (lesions) | 1850
Percent Diameter stenosis | 69.6 (15.4)

10. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: as for outcome 9
Time Frame: On day 0 after procedure
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: lesions
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1548
Number analyzed (lesions) | 1850
Percent Diameter stenosis | 23.6 (10.7)

11. Secondary Outcome: Percent Diameter Stenosis (%DS)
Description: as for outcome 9
Time Frame: At 8 months
Population: Eight-month follow-up angiograms for 1,309 lesions in 1,085 patients were assessed by the core laboratory.
Measure: Mean (Standard Deviation); unit: Percent Diameter stenosis
Units Other Than Participants: lesions
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1085
Number analyzed (lesions) | 1309
Percent Diameter stenosis | 26.1 (14.5)

12. Secondary Outcome: Acute Gain
Description: The acute gain was defined as the difference between post- and pre procedural minimal lumen diameter (MLD).
Time Frame: On day 0 after procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (95% Confidence Interval); unit: millimeters
Units Other Than Participants: lesions
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1548
Number analyzed (lesions) | 1850
millimeters
  In-stent (n=1845 lesions) | 1.769 [1.744 to 1.794]
  In-segment (n=1846 lesions) | 1.409 [1.383 to 1.436]

13. Secondary Outcome: Late Loss
Description: Proximal and distal late loss was calculated by [post-procedure minimum lumen diameter (MLD)] - [MLD at 8 months].
Time Frame: On day 0 after procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (95% Confidence Interval); unit: millimeters
Units Other Than Participants: lesions
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1548
Number analyzed (lesions) | 1850
millimeters
  In-stent (n=1303 lesions) | 0.219 [0.196 to 0.243]
  Proximal (n=1086 lesions) | 0.152 [0.125 to 0.178]
  Distal (n=1298 lesions) | 0.034 [0.012 to 0.055]
  In-segment (n=1308 lesions) | 0.128 [0.099 to 0.157]

14. Secondary Outcome: Net Gain
Description: Net Gain = Acute Gain - Late Loss, paired analysis only.
Time Frame: On day 0 after procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (95% Confidence Interval); unit: millimeters
Units Other Than Participants: lesions
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1548
Number analyzed (lesions) | 1850
millimeters
  In-stent (n=1300 lesions) | 1.536 [1.504 to 1.568]
  In-segment (n=1305 lesions) | 1.269 [1.235 to 1.302]

15. Secondary Outcome: Acute Success
Description: Acute Success: Procedural Success (Subject Level Analysis): Stent implant procedure was considered successful when all of the following criteria were met:
  * Stent was successfully delivered to the intended location
  * Stent was successfully deployed at the intended location
  * Stent delivery system was withdrawn without any issue Stent implantation procedure was considered successful in 99.94% of the stents. There was no stent adjudicated as procedure failure.
Time Frame: On day 0 (Immediately post-index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: percentage of stents
Units Other Than Participants: stents
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 2009
Number analyzed (stents) | 3104
percentage of stents
  Success | 99.94
  Unknown | 0.06

16. Secondary Outcome: Number of Participants With Any Death (Cardiac Death, Vascular Death, or Non-cardiovascular Death)
Description: All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in subjects with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
  • Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  • Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  • Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 47

17. Secondary Outcome: Number of Participants With Any Death (Cardiac Death, Vascular Death, or Non-cardiovascular Death)
Description: as for outcome 16
Time Frame: From 1 to 2 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 80

18. Secondary Outcome: Number of Participants With Any Death (Cardiac Death, Vascular Death, or Non-cardiovascular Death)
Description: as for outcome 16
Time Frame: From 2 years to 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 109

19. Secondary Outcome: Number of Participants With Myocardial Infarctions (MI)
Description: Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 17

20. Secondary Outcome: Number of Participants With Myocardial Infarctions (MI)
Description: as for outcome 19
Time Frame: From 1 year to 2 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 30

21. Secondary Outcome: Number of Participants With Myocardial Infarctions (MI)
Description: as for outcome 19
Time Frame: From 2 years to 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 33

22. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: Target Lesion Revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as clinically indicated [CI] or not clinically indicated by the investigator prior to repeat angiography. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement.
  The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the scaffold/stent.
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 72

23. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 22
Time Frame: From 1 year to 2 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 92

24. Secondary Outcome: Number of Participants With Target Lesion Revascularization (TLR)
Description: as for outcome 22
Time Frame: From 2 years to 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 104

25. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: Target Vessel Revascularization is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 113

26. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 25
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 146

27. Secondary Outcome: Number of Participants With Target Vessel Revascularization (TVR)
Description: as for outcome 25
Time Frame: From 2 Years to 3 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 168

28. Secondary Outcome: Number of Participants With Cardiac Death and All MI
Description: Cardiac death is defined as any death in which a cardiac cause cannot be excluded. (This includes but is not limited to acute myocardial infarction, cardiac perforation/pericardial tamponade, arrhythmia or conduction abnormality,cerebrovascular accident within 30 days of the procedure or cerebrovascular accident suspected of being related to the procedure, death due to complication of the procedure, including bleeding, vascular repair, transfusion reaction, or bypass surgery.)
  Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  -Non-Q wave MI: Elevation of CK levels to ≥ two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves.
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 31

29. Secondary Outcome: Number of Participants With Cardiac Death and All MI
Description: as for outcome 28
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 51

30. Secondary Outcome: Number of Participants With Cardiac Death and All MI
Description: as for outcome 28
Time Frame: From 2 Years to 3 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 56

31. Secondary Outcome: Number of Participants With Cardiac Death, All MI and Clinically-indicated Target Lesion Revascularization (CI-TLR)
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 87

32. Secondary Outcome: Number of Participants With Cardiac Death, All MI and Clinically-indicated Target Lesion Revascularization (CI-TLR)
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 120

33. Secondary Outcome: Number of Participants With Cardiac Death, All MI and Clinically-indicated Target Lesion Revascularization (CI-TLR)
Time Frame: From 2 Years to 3 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 133

34. Secondary Outcome: Number of Participants With Cardiac Death, Target Vessel Myocardial Infarction (TVMI) and TLR
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 96

35. Secondary Outcome: Number of Participants With Cardiac Death, Target Vessel Myocardial Infarction (TVMI) and TLR
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 125

36. Secondary Outcome: Number of Participants With Cardiac Death, Target Vessel Myocardial Infarction (TVMI) and TLR
Time Frame: From 2 Years to 3 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 140

37. Secondary Outcome: Number of Participants With Cardiac Death, All MI and Clinically-indicated Target Vessel Revascularization (CI-TVR)
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 122

38. Secondary Outcome: Number of Participants With Cardiac Death, All MI and Clinically-indicated Target Vessel Revascularization (CI-TVR)
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 163

39. Secondary Outcome: Number of Participants With Cardiac Death, All MI and Clinically-indicated Target Vessel Revascularization (CI-TVR)
Time Frame: From 2 Years to 3 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 184

40. Secondary Outcome: Number of Participants With All Deaths and All MI
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 61

41. Secondary Outcome: Number of Participants With All Deaths and All MI
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 105

42. Secondary Outcome: Number of Participants With All Deaths and All MI
Time Frame: From 2 Years to 3 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 134

43. Secondary Outcome: Number of Participants With All Deaths, All MI and All Revascularization
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 345

44. Secondary Outcome: Number of Participants With All Deaths, All MI and All Revascularization
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 449

45. Secondary Outcome: Number of Participants With All Deaths, All MI and All Revascularization
Time Frame: From 2 Years to 3 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 508

46. Secondary Outcome: Number of Participants With All Deaths, TVMI and TLR
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 126

47. Secondary Outcome: Number of Participants With All Deaths, TVMI and TLR
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 176

48. Secondary Outcome: Number of Participants With All Deaths, TVMI and TLR
Time Frame: From 2 Years to 3 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 214

49. Secondary Outcome: Number of Participants With All Deaths, TVMI and CI-TLR
Time Frame: Post Procedure to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1948
participants | 113

50. Secondary Outcome: Number of Participants With All Deaths, TVMI and CI-TLR
Time Frame: From 1 Year to 2 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1921
participants | 161

51. Secondary Outcome: Number of Participants With All Deaths, TVMI and CI-TLR
Time Frame: From 2 Years to 3 Years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Number; unit: participants
Arm/Group | XIENCE V / PROMUS Stent
Number analyzed (Participants) | 1890
participants | 196

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | XIENCE V / PROMUS Stent
All-Cause Mortality (participants affected / at risk) | 184/2009
Serious Adverse Events (participants affected / at risk) | 910/2009
Other Adverse Events (participants affected / at risk) | 116/2009
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE V / PROMUS Stent (N=2009)
Mild: bleeding that is not moderate nor severe (Blood and lymphatic system disorders) | 19
Moderate: bleeding that requires blood transfusion but does not result in hemodynamic compromise (Blood and lymphatic system disorders) | 21
Severe/Life Threatening (either intracranial hemorrhage or bleeding that causes hemodynamic compromi (Blood and lymphatic system disorders) | 19
Abnormal stress test (Cardiac disorders) | 9
Acute coronary syndrome (Cardiac disorders) | 18
Angina-equivalent symptoms (Cardiac disorders) | 108
Arrhythmia of unknown reason (Cardiac disorders) | 2
Atrial arrhythmia (Cardiac disorders) | 16
Cardiac arrest (Cardiac disorders) | 7
Cardiac: other (Cardiac disorders) | 3
Cardiomyopathy (Cardiac disorders) | 3
Cardiopulmonary arrest (Cardiac disorders) | 9
Conduction disorder (Cardiac disorders) | 17
Elevated cardiac enzymes (Cardiac disorders) | 4
Heart failure (Cardiac disorders) | 86
Hypertension (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 11
Palpitation (Cardiac disorders) | 4
Pericardial effusion (Cardiac disorders) | 1
Restenosis (Cardiac disorders) | 158
Stenosis (Cardiac disorders) | 244
Stent Thrombosis (Cardiac disorders) | 6
Tachycardia (Cardiac disorders) | 3
Tamponade (Cardiac disorders) | 1
Valve disorder (Cardiac disorders) | 10
Ventricular arrhythmia (Cardiac disorders) | 14
Biliary/liver disorder (Gastrointestinal disorders) | 26
Gastroesophageal reflux disease, diarrhea, nausea (Gastrointestinal disorders) | 21
Other gastro-intestinal symptoms (Gastrointestinal disorders) | 28
Pancreatic disorder (Gastrointestinal disorders) | 4
Abnormal Lab Test (Non-cardiac):Abnormal CBC with differentials (General disorders) | 4
Abnormal Lab Test (Non-cardiac):Abnormal liver enzymes (General disorders) | 1
Abnormal Lab Test (Non-cardiac):Abnormal other (General disorders) | 5
Contusion (General disorders) | 3
Death of unknown reason (General disorders) | 23
Eye/ear/nose/throat disorder (General disorders) | 23
Fall (General disorders) | 2
Fever (General disorders) | 3
Non cardiac chest pain (General disorders) | 0
General/Musculoskeletal/ Connective: Other (General disorders) | 29
Outcome to Death (General disorders) | 138
Weakness/fatigue (General disorders) | 3
Allergic Reaction to antiplatelet Agent (Immune system disorders) | 1
Allergic Reaction to contrast (Immune system disorders) | 3
Local infection (Infections and infestations) | 26
Systemic infection (Infections and infestations) | 16
Wound infection/abnormal healing (Infections and infestations) | 6
Diabetes mellitus (Metabolism and nutrition disorders) | 9
Hyper/hypoglycemia (Metabolism and nutrition disorders) | 1
Thyroid disorder (Metabolism and nutrition disorders) | 2
Ache/ myalgia/ pain (Musculoskeletal and connective tissue disorders) | 3
Bone or joint injury/disorder (Musculoskeletal and connective tissue disorders) | 42
Edema (Musculoskeletal and connective tissue disorders) | 3
Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15
Cancer and tumour: other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 100
Dizziness (Nervous system disorders) | 7
Headache/migraine (Nervous system disorders) | 1
Nerve/Psychiatric Disorders : Other (Nervous system disorders) | 9
Neuropathy (Nervous system disorders) | 2
Sleep disorder (Nervous system disorders) | 2
Stroke/CVA (Nervous system disorders) | 36
Syncope/fainting (Nervous system disorders) | 8
Genito-urinary and renal disorder (Renal and urinary disorders) | 40
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Chronic Obstructive Pulmonary Disease (COPD) (Respiratory, thoracic and mediastinal disorders) | 3
Interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 50
Respiratory System: other (Respiratory, thoracic and mediastinal disorders) | 9
Respiratory insufficiency/failure (Respiratory, thoracic and mediastinal disorders) | 5
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Rash/Urticaria (Skin and subcutaneous tissue disorders) | 2
skin/subcutaneous disorder: other (Skin and subcutaneous tissue disorders) | 4
Abrupt closure (Vascular disorders) | 1
Aneurysm (Vascular disorders) | 15
Dissection (Vascular disorders) | 2
Embolism (Vascular disorders) | 4
Hematoma (Vascular disorders) | 7
Ischemia (Vascular disorders) | 10
No/slow reflow (Vascular disorders) | 2
Occlusion (Vascular disorders) | 14
Perforation (Vascular disorders) | 3
Peripheral arterial disease (Vascular disorders) | 35
Peripheral vascular disease (PVD) (Vascular disorders) | 0
Spasm (Vascular disorders) | 1
Thrombosis - non stent (Vascular disorders) | 6
Vascular: other (Vascular disorders) | 17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XIENCE V / PROMUS Stent (N=2009)
Mild: bleeding that is not moderate nor severe (Blood and lymphatic system disorders) | 1 — Bleeding
Moderate: bleeding that requires blood transfusion but does not result in hemodynamic compromise (Blood and lymphatic system disorders) | 1 — Bleeding
Abnormal stress test (Cardiac disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 3
Angina-equivalent symptoms (Cardiac disorders) | 23
Arrhythmia of unknown reason (Cardiac disorders) | 1
Cardiopulmonary arrest (Cardiac disorders) | 6
Conduction disorder (Cardiac disorders) | 1
Elevated cardiac enzymes (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 6
Myocardial infarction (Cardiac disorders) | 2
Palpitation (Cardiac disorders) | 1
Restenosis (Cardiac disorders) | 44
Stenosis (Cardiac disorders) | 20
Stent Thrombosis (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Ventricular arrhythmia (Cardiac disorders) | 6
Biliary/liver disorder (Gastrointestinal disorders) | 1
Gastro-intestinal disorder (e.g. GERD, diarrhea, nausea) (Gastrointestinal disorders) | 1
Non cardiac chest pain (General disorders) | 0
General/Musculoskeletal/ Connective : Other (General disorders) | 4 — Except bone or joint injury/disorder and Non cardiac chest pain.
Allergic Reaction:To antiplatelet Agent (Immune system disorders) | 1 — Allergic Reaction
Wound infection/abnormal healing (Infections and infestations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 — Metabolism/endocrine
Hyper/hypoglycemia (Metabolism and nutrition disorders) | 1 — Metabolism/endocrine
Bone or joint injury/disorder (Musculoskeletal and connective tissue disorders) | 4 — Systemic/musculoskeletal/connective tissue disorder
Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Cancer and Tumor
Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 — Cancer and Tumor
Nerve/psychiatric disorders : Other (Nervous system disorders) | 1
Genito-urinary and renal disorder (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0
Respiratory/Pulmonary disorders : Other (Respiratory, thoracic and mediastinal disorders) | 1
Dissection (Vascular disorders) | 1
Ischemia (Vascular disorders) | 4
Jailing of side branch (Vascular disorders) | 1
No/slow reflow (Vascular disorders) | 1
Perforation (Vascular disorders) | 1
Peripheral artery disease (PAD) (Vascular disorders) | 2
Spasm (Vascular disorders) | 2
Thrombosis - non stent (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days